CLINICAL TRIAL: NCT07037329
Title: To Determine the Effectiveness of TENS vs EMS on Hemodynamics Parameters of Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1012
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Electrical Nerve Stimulation (TENS) (Experimental)
  Interventions: Diagnostic Test: Transcutaneous Electrical Nerve Stimulation (TENS)
- Electrical Muscle Stimulation (EMS) (Experimental)
  Interventions: Diagnostic Test: Electrical Muscle Stimulation (EMS)

INTERVENTIONS:
Diagnostic Test: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS is a non-invasive electrotherapy technique used to manage pain and modulate physiological responses such as blood pressure. In this study, patients in Group 1 received TENS therapy as the primary intervention.
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)
Diagnostic Test: Electrical Muscle Stimulation (EMS) — EMS is a form of electrotherapy that causes muscle contractions through electrical impulses delivered via surface electrodes. In this study, patients in Group 2 received EMS therapy to investigate its effect on hemodynamic parameters in individuals with hypertension.
  Arms: Electrical Muscle Stimulation (EMS)

SUMMARY:
This study aimed to evaluate the comparative effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS) and Electrical Muscle Stimulation (EMS) on hemodynamic parameters in patients with hypertension. A total of 42 hypertensive patients were randomly divided into two equal groups: Group A received TENS, and Group B received EMS, over a period of four weeks. Pre- and post-treatment measurements of systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate (HR) were recorded. Results showed that both TENS and EMS produced significant improvements in all parameters within their respective groups.

DETAILED DESCRIPTION:
However, the TENS group demonstrated a greater reduction in SBP and DBP, while the EMS group showed better improvement in heart rate control. The findings suggest that both treatments are effective non-pharmacological options for managing hypertension, with TENS being more effective overall in lowering blood pressure. These modalities may offer supportive benefits in long-term hypertension management strategies.

ELIGIBILITY:
Inclusion Criteria:

* (25-60 years) including both male and female
* Patients clinically diagnosed with primary (essential) hypertension.
* Blood pressure ranging from 140/90 mmHg to 160/100 mmHg (Stage 1 to early Stage 2 hypertension).
* Participants who are not currently on intensive antihypertensive therapy or are on a stable dose of medication.
* Willingness to participate voluntarily and provide written informed consent.
* Patients who are not involved in any physical activity.
* Participants who are overweight according to normal BMI.

Exclusion Criteria:

* Secondary hypertension due to renal, endocrine, or other systemic causes. Individuals with pacemakers, implanted defibrillators, or other electronic medical devices.
* Patients with severe cardiovascular conditions, such as recent myocardial infarction, heart failure, or arrhythmias.

History of seizure disorders or epilepsy. Cancer Patients

* Presence of skin lesions, open wounds, or infections at the site of electrode placement.
* Patients undergoing physiotherapy or electrical therapy elsewhere during the study period.
* Individuals with known neurological or musculoskeletal disorders that could interfere with EMS or TENS effectiveness

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
SF-36 Health Survey (Optional for Quality of Life) | 6 Month
  Measures general health status and quality of life 36 items grouped into 8 domains (e.g., physical functioning, general health)
  Each domain scored from 0 (worst) to 100 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Yasin Poly Clinic, Behria town Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No